CLINICAL TRIAL: NCT01869985
Title: A Randomized, Open-label, Single Dose, 3-sequence and 3-period Partial Replicated Crossover Clinical Study to Compare Pharmacokinectic Characteristics of Eperisone Hydrochloride and Aceclofenac With HCP1104 Treatment to Those of Co-administration of Eperisone Hydrochloride 50mg Tablet and Aceclofenac 100mg Tablet in Healthy Adult Male Volunteers
Brief Title: Partial Replicated Crossover Clinical Study to Compare Pharmacokinectic Characteristics of Eperisone Hydrochloride and Aceclofenac With HCP1104 Treatment to Those of Co-administration of Eperisone Hydrochloride 50mg Tablet and Aceclofenac 100mg Tablet in Healthy Adult Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-EPAC-102
Record Dates: First submitted 2013-06-03; First posted 2013-06-05 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Healthy
Keywords: HCP1104; Eperisone Hydrochloride; Aceclofenac
MeSH Terms: interventions — aceclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HCP1104 (Experimental): HCP1104
  Interventions: Drug: HCP1104 / Mulex Tab. and Airtal Tab.
- Mulex Tab. and Airtal Tab. (Active Comparator): Eperisone Hydrochloride and Aceclofenac
  Interventions: Drug: HCP1104 / Mulex Tab. and Airtal Tab.

INTERVENTIONS:
Drug: HCP1104 / Mulex Tab. and Airtal Tab. — HCP1104 / Eperisone plus Aceclofenac

SUMMARY:
The purpose of this study is to evaluate pharmacokinetics and safety after oral administration of HCP1104 and Eperisone Hydrochloride plus Aceclofenac.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate pharmacokinetics and safety after oral administration of HCP1104 and Eperisone Hydrochloride plus Aceclofenac.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers, age between 20 and 45
* BMI of >20kg/m2 and <28kg/m2 subject
* Informed of the investigational nature of this study and voluntarily agree to participate in this study

Exclusion Criteria:

* Use of any prescription medication within 14 days prior to Day 1
* Use of any medication within 7 days prior to Day 1
* Participation in another clinical study within 60 days prior to start of study drug administration

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-08; Primary Completion 2013-09 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Area Under Curve(AUC) last | 0, 20, 40min, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24h hours post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea